CLINICAL TRIAL: NCT06778564
Title: Augmentation With Cannabidiol in First Episode Psychosis: a Double-blind, Randomised Controlled Trial
Brief Title: Stratification and Treatment in Early Psychosis Study - ENHANCE
Acronym: STEP-ENHANCE
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Wellcome Trust (Other); Cambridge Cognition Ltd (Industry); Cambridgeshire and Peterborough NHS Foundation Trust (Other); Oxford Health NHS Foundation Trust (Other Government); West London NHS Trust (Other); Charite University, Berlin, Germany (Other); University of Cologne (Other); Ludwig-Maximilians - University of Munich (Other); The Sheba Fund for Health Services and Research (Unknown); Shalvata Mental Health Center (Other); Geha Mental Health Center (Other); Amsterdam University Medical Center (Other); Hospital General Universitario Gregorio Marañon (Other); National and Kapodistrian University of Athens (Other); Medical University of Vienna (Other); Hospitales Universitarios Virgen del Rocío (Other); University of Campania Luigi Vanvitelli (Other); Psychiatric University Hospital, Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PID-17638; 2025-521929-32-00 (EU CTIS Number); 1008451 (Other: HRA UK -IRAS)
Record Dates: First submitted 2024-12-12; First posted 2025-01-16 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2024-12

CONDITIONS: Psychosis; First Episode Psychosis; Psychotic Disorders; Psychotic Episode
Keywords: Cannabidiol; first episode psychosis
MeSH Terms: conditions — Psychotic Disorders | interventions — Solutions

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled
Who Masked: Participant, Outcomes Assessor
Masking Description: Double blind - CBD and placebo will have an identical appearance, taste and texture.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cannabidiol (CBD) (Experimental): Participants in this arm will receive Cannabidiol (CBD) for 6 weeks.
  Interventions: Drug: CBD 100 mg/mL Oral Solution
- Placebo (Placebo Comparator): Participants in this arm will receive placebo for 6 weeks.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CBD 100 mg/mL Oral Solution — Daily dose 1000mg, taken as 500mg (5ml) b.i.d for 6 weeks. For participants with a weight lower than 50 kg, the dose is to be adjusted to 20 mg/kg/day divided over 2 intakes of 10 mg/kg/day, for a period of 6 weeks
  Arms: Cannabidiol (CBD)
Other: Placebo — 5ml b.i.d for 6 weeks; For participants with a weight lower than 50 kg, the dose is to be adjusted to 20 mg/kg/day divided over 2 intakes of 10 mg/kg/day, for a period of 6 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is:

* To investigate whether the response to antipsychotic treatment can be enhanced by adding cannabidiol (CBD) to the existing treatment, compared to placebo, in participants with a first episode of psychosis, who have had a suboptimal or no response to their first antipsychotic treatment.
* To confirm the safety of CBD in people with psychosis.

The study is a randomized, double-blind, placebo-controlled, multi-centre, clinical trial. Individuals with a diagnosis of first-episode psychosis, who have had a suboptimal or no response to their first antipsychotic treatment will be recruited. These participants are randomised to treatment with CBD oral solution 500mg twice daily, or a matching placebo for 6 weeks, as an adjunct to their existing antipsychotic treatment. By using a battery of clinical outcome assessments, the trial will also assess several biomarkers to determine if they can be used to predict clinical outcomes and response to treatment with CBD. Biomarkers are being assessed as an exploratory outcome measure. Participants will be invited to provide blood and stool samples, and may be asked to complete neuroimaging assessments at certain eligible sites.

ELIGIBILITY:
Inclusion criteria:

1. The participant is 16 to 40 years of age, willing and able to provide written informed consent/assent.
2. The participant is currently being treated with an antipsychotic for at least 3 weeks but no longer than 16 weeks.
3. The participant should be receiving at least the minimum dose of this antipsychotic for FEP according to modified Maudsley guidelines, as listed in Appendix B. The clinician should judge the participant to be a non-responder to this treatment and that increasing the dose further is unacceptable to the clinician and/or participant.
4. The compliance score associated with this antipsychotic medication is 4 or more on the Clinician Rating Scale (CRS).
5. The participant meets DSM-5 criteria for schizophrenia, schizoaffective disorder or schizophreniform disorder, as confirmed through the SCID-5-RV.
6. The participant does not meet modified Andreasen criteria for symptomatic remission (time requirement does not apply).
7. Participants of childbearing potential (*) must be willing to ensure that they use highly effective contraception during the trial and as per the requirements in the protocol**.
8. In the Investigator's opinion, is able and willing to comply with all trial requirements.
9. Willing to allow their General Practitioner and/or consultant, if required by local guidelines/regulations, to be notified of participation in the trial.
10. For participants who take part in the optional MRI scans: they must be eligible for MRI scanning as per local requirements, for example concerning e.g. implants, braces etc.

There is inadequate information on the effects of cannabidiol on the foetus in humans. Participants of childbearing potential* should use a highly effective method of contraception** for the duration of the trial and for 3 months after the last time the trial intervention was used.

*A person is considered of childbearing potential, i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause.

** Methods that can achieve a failure rate of less than 1% per year when used consistently and correctly are considered as highly effective birth control methods. Such methods include: 1) combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral; intravaginal; transdermal); 2) progestogen-only hormonal contraception associated with inhibition of ovulation (oral; injectable; implantable); 3) intrauterine device (IUD); 4) intrauterine hormone-releasing system (IUS); 5) bilateral tubal occlusion; 6) vasectomised partner; 7) sexual abstinence (abstinence should only be used as a contraceptive method if it is in line with the participants' usual and preferred lifestyle).

Periodic abstinence (calendar, symptothermal, post-ovulation methods) is not an acceptable method of contraception. The participant agrees to use an acceptable method of contraception* for the duration of the study and for 3 months after any study drug administration, unless surgically sterile or postmenopausal (no menses for 12 months without an alternative medical cause).

The age range for eligibility has been applied as this corresponds to the usual age range for first episode psychosis; individual cases outside of this age range may have a different aetiology and/or prognosis which could impact on the study outcomes.

Exclusion criteria:

1. Having been previously treated with a different antipsychotic (to the current one) at an adequate dose* for 4 weeks or longer.
2. Current or previous treatment with clozapine and/or current treatment with sodium valproate, valproate semisodium, or clobazam. In cases of current use of these medicines, participation is only permitted if they can and will be discontinued or switched to a suitable alternative medication prior to randomisation.
3. Hypersensitivity to the active substance, sesame oil, sesame seed or any of the excipients of the intervention.
4. Known hepatic insufficiency and/or transaminase elevations levels exceeding the upper limit of normal 2 times or more and bilirubin greater than 1.5 times the upper limit of normal.
5. Previous neurosurgery or neurological disorder, including epilepsy, which may affect the study procedures**.
6. IQ <70.
7. Pregnancy or breastfeeding.
8. The patient has a current diagnosis of 'Substance or medication induced psychotic disorder' or 'Psychotic disorder due to another medical condition' as determined through the SCID-5-RV.
9. Current active suicidal ideation within the last 2 weeks, defined as a score of 1 or higher on CDSS question 8, followed by an assessment by the treating clinician who determines it is not safe for the patient to participate in the study***.
10. Meeting DSM-V criteria for substance use disorder, with the exception of nicotine use disorder (mild, moderate, and severe allowed). Mild cannabis use disorder is allowed (i.e. can meet up to but no more than 3 criteria on the SCID) as long as the subject patient has not consumed cannabis on average more than three times a week in the past 30 days. Mild alcohol use disorder is also allowed.
11. Patient has participated in another clinical trial in which they received an experimental or investigational drug or agent within 3 months before Visit 0. Patients who have participated in Type A studies (e.g. trials of standard and within-label treatments including antipsychotic medication) or non CTIMP studies (e.g. studies of exercise therapy) must have completed the intervention but may be included if permitted by the protocol of the other trial.
12. The participant refuses any mandatory safety checks during the trial, specifically, refusal of: urine pregnancy test (those of child-bearing potential only); safety blood test; reporting of adverse events; and assessment of suicidality.
13. Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.

    * Adequate doses are provided in Appendix B. **Minor neurological disorders such as migraine, other minor headache disorders, sleep disorders or nerve palsies which are unlikely to affect study outcomes including neuroimaging measures are permitted.

      * The decision to include the patient is at clinician's discretion. The clinician can conclude that it is safe for the patient to participate after the patient is evaluated, in which case this exclusion criterion does not apply and the patient can participate. Either way, the treating clinician needs to record his/her evaluation of suicidal risk in the source documentation or medical file, including his/her considerations, and notify the site PI of the decision.

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 250 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Change in Positive and Negative Syndrome Scale (PANSS) total score | 6 weeks
  Change in Positive and Negative Syndrome Scale (PANSS) total score from baseline to 6 weeks. The minimum value is 1 and the maximum value is 7 for each item of the scale.
  1. A patient meets remission criteria if none of the following items score a 4 or higher: P1, P2, P3, N1, N4, N6, G5 and G9.
  2. A patient does not meet remission criteria if one or more of these items score a 4 or higher.

SECONDARY OUTCOMES:
Change in symptoms (sub-scale scores) | from baseline to 6 weeks and 58weeks
  Change in scores on the PANSS positive, negative and general symptom subscales from baseline to 6 weeks and 58 weeks (if participants consent to the optional 12 months long-term follow-up period).
Symptomatic remission | 6 weeks and 58weeks
  Symptomatic remission after 6 weeks and 58 weeks (if participants consent to the optional 12 months long-term follow-up period as measured using the PANSS, defined using Andreasen (2005) remission criteria.
  Andreasen, N. C., Carpenter, W. T., Jr, Kane, J. M., Lasser, R. A., Marder, S. R., & Weinberger, D. R. (2005). Remission in schizophrenia: proposed criteria and rationale for consensus. The American journal of psychiatry, 162(3), 441-449. https://doi.org/10.1176/appi.ajp.162.3.441
Change in overall clinical impression | from baseline to 6 weeks and 58weeks
  Change in overall clinical impression, assessed through Clinical Global Impression of Improvement and Severity (CGI-I/S) scales from baseline to 6 weeks and 58 weeks (if participant consent to the optional 12 months long-term follow-up period).
Change in functioning | from baseline to 6 weeks and 58weeks
  Change in functioning, assessed through Social and Occupational Function Scale (SOFAS) from baseline to 6 weeks and 58 weeks (if participants consent to the optional 12 months long-term follow-up period).
  Score range 1-100, the higher score means the better function
Change in functioning | from baseline to 6 weeks and 58weeks
  Change in functioning, assessed through Functional Remission of General Schizophrenia scale (FROGS) from baseline to 6 weeks and 58 weeks (if participants consent to the optional 12 months long-term follow-up period).
  Scale range for each item: Do not do=1; Do partially=2; Do a significant part=3; Do almost all the activity=4; Do perfectly =5. The higher score means better functioning.
Change in functioning | from baseline to 6 weeks and 58weeks
  Change in functioning, assessed through Global Functioning Social and Role scales (GF:S, GF:R) from baseline to 6 weeks and 58 weeks (if participants consent to the optional 12 months long-term follow-up period).
  Scale range 1-100;
  1. Different reference period at follow-ups: time since last visit
  2. Rate only at baseline At follow-up, the higher score during past observation period can only be above but not below the current score at the last visit (i.e. if lower, the current score of last visit defines score during past observation (usually last 3 months)). The lowest score during past observation period can only be below but not above the current score at the last visit.
Change in cognitive functioning | from baseline to 6 weeks
  Change in cognitive functioning as assessed through the PsyCog battery from baseline to 6 weeks.
  PsyCog comprises four tests that were chosen from the larger CANTAB battery to assess the key cognitive deficits associated with psychosis, including::
  * Paired Associates Learning (PAL): key measures including PAL total errors adjusted (score range 0-70; lower is better) and PAL first attempt memory score (score range 0-20; higher is better)
  * Rapid Visual Information Processing (RVP): key measures including RVP A' (score range 0-1; higher is better) and RVP median response latency(ms) (score range 100-1900; lower is better)
  * Emotion Recognition Task (ERT): key measures including ERT overall median reaction time (ms) (score range 100-00; lower is better) and ERT total hits (score range 0-48; higher is better)
  * Spatial Span (SSP): key measures including SSP forward span length (score range 3-9; higher is better) and SSP reserve span length (score range 3-9; higher is better)
Change in quality of life | from baseline to 6 weeks and 58weeks
  Change in quality of life, assessed using the EQ-5D three-level version (EQ-5D-3L) from baseline to 6 weeks and 58 weeks (if participants consent to the optional 12 months long-term follow-up period). It includes five dimensions-MOBILITY, SELF-CARE, USUAL ACTIVITIES, PAIN /DISCOMFORT and ANXIETY / DEPRESSION. Each dimension has three levels: no problems, some problems, extreme problems (labelled1-3). The respondent is asked to indicate his / her health state by checking the box against the most appropriate statement in each of the five dimensions.
  The EQ VAS records the respondent's self-rated health on a vertical VAS where the endpoints are labelled 'The best health you can imagine' and 'The worst health you can imagine'. This information can be used as a quantitative measure of health outcome as judged by the individual respondents.
Change in quality of life | from baseline to 6 weeks and 58weeks
  Change in quality of life, assessed using the World Health Organization Quality-of-Life Scale (WHOQOL-BREF) from baseline to 6 weeks and 58 weeks (if participants consent to the optional 12 months long-term follow-up period).
  The WHOQOL-BREF is a 26-item instrument consisting of four domains: physical health (7 items), psychological health (6 items), social relationships (3 items), and environmental health (8 items); it also contains QOL and general health items. Each individual item of the WHOQOL-BREF is scored from 1 to 5 on a response scale, which is stipulated as a five-point ordinal scale.
Acceptability of CBD treatment | 6 weeks
  Acceptability of CBD treatment, measured through all-cause discontinuation over 6 weeks
Incidence of adverse events | 6 weeks and 30 days post treatment
  Incidence of adverse events, measured through Glasgow Antipsychotic Side-effect Scale (GASS) over 6 weeks. Spontaneous adverse event reporting is until 30 days after the study intervention has been discontinued.
Changes in measuring the severity of anxiety and depression symptoms | from baseline to 6 weeks
  Measure the severity of anxiety symptoms via Hamilton Anxiety Scale (HAM-A) from baseline to 6weeks.
  Each item is scored on a scale of 0 (not present) to 4 (severe), with a total score range of 0-56, where <17 indicates mild severity, 18-24 mild to moderate severity and 25-30 moderate to severe.
Changes in measuring the severity of anxiety and depression symptoms | from baseline to 6 weeks
  Measure the severity of anxiety symptoms via the Overall Anxiety Severity and Impairment Scale (OASIS) from baseline to 6weeks.
  It consists of five items that measure the frequency and severity of anxiety, as well as level of avoidance, work/school/home interference, and social interference associated with anxiety. Respondents select among five different response options for each item, which are coded 0-4 and summed to obtain a total score. Score range is 0-20. The lower score is better in symptoms.
Changes in measuring the depression symptoms | from baseline to 6 weeks
  Measure the depression in schizophrenia without overlap with negative symptoms and extrapyramidal symptoms by using the Calgary Depression Scale for schizophrenia (CDSS) from baseline to 6weeks.
  it includes 9 items in the scale. All ratings of the items are defined according to operational criteria from 0-3. The CDSS depression score is obtained by adding each of the item scores. Score range is 0-27, which is the lower score is better.
Changes in biomarkers that occur in relation to symptomatic improvement with adjunctive cannabidiol compared to placebo. | baseline and 6 weeks
  Measure the neuroimaging (Magnetic resonance imaging (MRI)) from baseline to 6 weeks if participant consents to it.
  The Magnetic resonance imaging (MRI) scan includes:
  T1 - brain structure T2 FLAIR - brain structure / clinical reporting Neuromelanin sensitive MRI - neuromelanin content of substantial nigra (proxy of dopamine activity) Magnetic Resonance Spectroscopy of the anterior cingulate cortex - metabolites e.g. glutamate Resting state fMRI - bold activation during "rest" or free mind wandering
Changes in biomarkers that occur in relation to symptomatic improvement with adjunctive cannabidiol compared to placebo. | baseline and 6 weeks
  Measure the microbiome samples from baseline to 6 weeks if participant consents to it.
  The gut-microbiome (the microorganisms e.g. bacteria, normally found in participant's gut) is likely to be at play in determining whether participant respond or experience side effects from CBD.
  Two tubes of stool samples to be collected at two time points(baseline and week 6) if participant consent to it.
Changes in biomarkers that occur in relation to symptomatic improvement with adjunctive cannabidiol compared to placebo. | from baseline to 6 weeks
  Measure the blood samples for central lab assessment including (Epi)genetics, proteomics, inflammation, metabolomics, Redox markers from baseline to 6 weeks if participant consents to it.

OTHER OUTCOMES:
Change in overall patient impression of severity and improvement | from baseline to 6 weeks and 58weeks
  Change in overall patient impression, assessed through Patient Global Impression of Improvement and Severity (PGI-I/S) scales from baseline to 6 weeks and 58 weeks (if participant consents to the optional 12 months long-term follow-up period) The Patient Global Impression of Improvement (PGI-I) is a single question asking the patient to rate how their psychotic symptoms is now compared to the previous study visit on a scale of 1. very much better to 7. very much worse. The lower score is better in symptoms' improvement.
  The Patient Global Impression of Severity (PGI-S) is a single question asking the patient to rate how their psychotic symptoms is now on a scale of 1. not present to 7. very severe. The lower score is better in symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Philip McGuire, PhD MD, Principal Investigator — University of Oxford
Locations (17):
- MedUni Vienna, Vienna, Austria
- Germany (4):
  - University of Augsburg, Augsburg
  - Charité Universitätsmedizin, Berlin
  - University Hospital Cologne, Cologne
  - Ludwig-Maximilian-University Munich, Munich
- National and Kapodistrian University of Athens, Athens, Greece
- Israel (3):
  - Shalvata Mental Health Center, Hod HaSharon
  - Geha Mental Health Center, Petah Tikva
  - Sheba Medical Centre, Ramat Gan
- University of Campania 'Luigi Vanvitelli', Napoli, Italy
- Stichting Amsterdam UMC, Amsterdam, Netherlands
- Spain (2):
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Virgen del Rocío, Seville
- Psychiatric University Hospital (PUK), Zurich, Zurich, Switzerland
- United Kingdom (3):
  - Cambridgeshire and Peterborough NHS Foundation Trust, Cambridge
  - West London NHS Trust, London
  - Oxford Health NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: Yes
Please contact the sponsor, who will provide instructions for submitting a data request. All data can be requested, regardless of the location of the requesting party.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data and supporting documents will become available once the primary papers are available in the scientific domain.
Access Criteria: These will be provided by the sponsor to the requesting party.